CLINICAL TRIAL: NCT00003575
Title: A Randomized Pre-Phase II Trial of Interleukin-2, Interleukin-12, or No Additional Therapy Following Response to Ifosfamide/Etoposide Chemotherapy for Refractory HIV-Associated Non-Hodgkin's Lymphoma
Brief Title: Interleukin-12 Following Chemotherapy in Treating Patients With Refractory HIV-Associated Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02276; AMC-008; CDR0000066642 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 1999-11-01; First posted 2004-05-20 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2002-10

CONDITIONS: Lymphoma
Keywords: AIDS-related peripheral/systemic lymphoma; AIDS-related diffuse large cell lymphoma; AIDS-related immunoblastic large cell lymphoma; AIDS-related small noncleaved cell lymphoma
MeSH Terms: conditions — Lymphoma | interventions — Filgrastim; Interleukin-12 Subunit p35; Etoposide; Ifosfamide

ARMS (1):
- Arm I (Experimental): All patients receive ifosfamide IV by continuous infusion for 2 days, etoposide IV over 2 hours daily on days 1 and 2, and filgrastim (G-CSF) subcutaneously (SC) daily on days 4-13. Courses are repeated every 21 days. Patients who have complete or partial remission after a minimum of 4 courses of chemotherapy receive maintenance therapy consisting of interleukin-12 SC twice weekly beginning on day 28 of the final chemotherapy course and continuing for 6 months or until disease progression. All patients also receive combination antiretroviral therapy during study.
  Interventions: Biological: filgrastim; Biological: recombinant interleukin-12; Drug: etoposide; Drug: ifosfamide

INTERVENTIONS:
Biological: filgrastim
Biological: recombinant interleukin-12
Drug: etoposide
Drug: ifosfamide

SUMMARY:
Phase II trial to compare the effectiveness of interleukin-12 following chemotherapy in treating patients who have refractory HIV-associated non-Hodgkin's lymphoma. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Interleukin-12 may kill tumor cells by stopping blood flow to the tumor and by stimulating a person' white blood cells to kill cancer cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the efficacy of interleukin-12 (IL-12) by evaluating its effect on remission duration after response to second line chemotherapy with ifosfamide and etoposide in patients with HIV-associated non-Hodgkin's lymphoma.

II. Determine the safety of IL-12 when administered as maintenance therapy in these patients.

III. Evaluate overall survival of this patient population. IV. Evaluate serum and tissue cytokine levels in these patients. V. Evaluate the effect of IL-12 on HIV viral load and on functional T-cell assays in these patients.

VI. Evaluate the effect of IL-12 on Epstein-Barr Virus (EBV) viral load in these patients.

OUTLINE: This is an open label study.

All patients receive ifosfamide IV by continuous infusion for 2 days, etoposide IV over 2 hours daily on days 1 and 2, and filgrastim (G-CSF) subcutaneously (SC) daily on days 4-13. Courses are repeated every 21 days. Patients who have complete or partial remission after a minimum of 4 courses of chemotherapy receive maintenance therapy consisting of interleukin-12 SC twice weekly beginning on day 28 of the final chemotherapy course and continuing for 6 months or until disease progression. All patients also receive combination antiretroviral therapy during study.

Patients are followed every month for one year, then every 2 months thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* HIV-infected patients with histologically or cytologically proven intermediate grade large cell lymphoma; high grade large cell immunoblastic lymphoma; or high grade small noncleaved cell lymphoma who have either failed to respond to or relapsed following first line combination chemotherapy
* Bidimensionally measurable disease
* No CNS lymphoma (parenchymal brain or spinal cord tumor)
* No meningeal lymphoma
* A new classification scheme for adult non-Hodgkin's lymphoma has been adopted by PDQ. The terminology of "indolent" or "aggressive" lymphoma will replace the former terminology of "low", "intermediate", or "high" grade lymphoma. However, this protocol uses the former terminology.

PATIENT CHARACTERISTICS:

* Age: 18 to 70
* Performance status: Karnofsky 60-100%
* Absolute neutrophil count at least 1,000/mm3
* Platelet count greater than 75,000/mm3
* Hematologic criteria not applicable if abnormal functions are attributable to lymphomatous infiltration of bone marrow or liver
* Bilirubin less than 2.0 mg/dL, except in patients receiving indinavir who have isolated hyperbilirubinemia
* Transaminases less than 5 times upper limit of normal
* Hepatic criteria not applicable if abnormal functions are attributable to lymphomatous infiltration of bone marrow or liver
* Creatinine clearance greater than 60 mL/min
* No other prior or concurrent malignancy except carcinoma in situ of the cervix or nonmetastatic nonmelanomatous skin cancer
* No acute active opportunistic infection requiring antibiotic treatment Patients with Mycobacterium avium complex allowed
* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* At least 2 weeks since prior immunomodulating agents
* Concurrent filgrastim (G-CSF) allowed
* Concurrent epoetin alfa allowed
* Concurrent antibiotics may be given if clinically indicated during study
* No more than 2 prior standard treatment regimens for non-Hodgkin's lymphoma
* No concurrent systemic corticosteroids
* Concurrent topical and/or oral antifungal agents permitted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1999-01; Primary Completion 2002-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence D. Kaplan, MD, Study Chair — University of California, San Francisco
Locations (10):
- United States (10):
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - San Francisco General Hospital Medical Center, San Francisco, California
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Robert H. Lurie Comprehensive Cancer Center, Northwestern University, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - University Hospital/New Jersey Cancer Center, Newark, New Jersey
  - NYU School of Medicine's Kaplan Comprehensive Cancer Center, New York, New York
  - Memorial Sloan-Kettering Cancer Center, New York, New York
  - Mount Sinai School of Medicine, New York, New York
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio